CLINICAL TRIAL: NCT06853119
Title: Study on Brain Function and Structural Changes in Patients with Trigeminal Neuralgia Based on Magnetic Resonance Imaging.
Brief Title: Magnetic Resonance Imaging in Patients with Trigeminal Neuralgia
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Professor, Tongji Hospital
Other Study IDs: 2024S240
Record Dates: First submitted 2025-02-15; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Trigeminal Neuralgia (TN)
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Trigeminal Neuralgia Group: Patients who were diagnosed with trigeminal neuralgia (TN) according to the International Classification of Headache Disorders (ICHD) and were intolerant or ineffective to the preoperative treatment of carbamazepine or ocasepine, requiring the treatment of percutaneous balloon compression (PBC)
- Health Control Group: Healthy controls matched by age, sex, etc

SUMMARY:
This study intends to use MRI technology to analyze the dynamic changes and microstructure changes of the brain network in patients with trigeminal neuralgia, evaluate the blood-brain barrier and water exchange rate, and further analyze their correlation with clinical indicators, so as to explore the changes in brain structural plasticity and potential neural mechanisms

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis was TN according to the ICHD.
* Patients requiring surgical treatment due to ineffective or intolerant treatment with carbamazepine or oxasepine before operation;
* First surgical treatment;
* Right-handed dominant;
* There was no significant loss of sensation

Exclusion Criteria:

* Secondary TN;
* Associated with other types of chronic pain or neuropsychiatric disorders;
* History of head trauma or stroke or cerebrovascular ischemia;
* History of microvascular decompression or other treatments (gamma knife radiosurgery, etc.);
* Unable to cooperate independently;
* Contraindications, such as uncontrolled infection, coagulopathy, etc.;
* MRIcontraindications (e.g., pacemaker, claustrophobia, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with TN undergoing PBC and healthy controls matched by age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Scanning sequence of magnetic resonance imaging (MRI) | Preoperative routine MRI examination
  such as 3D-T1, 3D-T2, BOLD-functional MRI (fMRI), diffusion weighted imaging (DWI) (Multiple b values, such as 0,1000,2000), diffusion-prepared, arterial spin labeling (DP-ASL), Meningeal lymphatic sequence (3D T2-FLAIR ).

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | Baseline, until to discharge (an average of 3 days), 3 months after surgery
  The BPI is divided into two parts, one of which assesses pain severity on a scale of 0 to 10, where 0 means "no pain" and 10 means "most severe pain." The other assessed the extent to which pain interfered with daily activities, including seven areas of general activity, mood, ability to walk, normal work (including housework), relationships, sleep, and enjoyment of life, with 0 being "no impact" and 10 being "significant impact."
Simplified McGill pain questionnaire (SF-MPQ) | Baseline, 3 months after surgery
  The scale consisted of two subscales with 11 pain description items and 4 emotional assessment items [pain-free (0), mild (1), moderate (2), severe (3)], and a visual analog scale (VAS) [0-10, painless (0), severe pain (10)] was added to assess pain intensity.
Douleur Neuropathique 4 Questions (DN4) | Baseline, 3 months after surgery
  The scale contains 10 items, divided into two parts: Symptom description (7 items) : covers burning pain, cold pain, electric shock pain, tingling pain, acupuncture pain, numbness, and pruritus. Clinical examination (3 items) : Includes loss of touch, loss of tingling, and whether rubbing in the pain area induces or worsens pain. "Yes" scores 1 point for each item, "no" scores 0 points, total score ≥4 points can be diagnosed as neuropathic pain
Beck Depression Inventory (BDI) | Baseline, 3 months after surgery
  BDI consists of 21 items, each corresponding to a common depressive symptom, such as sadness, insomnia, fatigue and feelings of worthlessness. Each item has four options, representing the severity of symptoms, on a scale of 0 (no symptoms) to 3 (severe symptoms). The overall score ranges from 0 to 63, with the higher the score, the more severe the depressive symptoms.
Beck Anxiety Inventory (BPI) | Baseline, 3 months after surgery
  BAI consists of 21 items, each describing an anxiety-related symptom, and subjects are required to choose the answer that best fits their situation based on their feelings in the past week. A 4-level scoring method was adopted:
  0: None
  1. Mild, not much bother
  2. Moderate, uncomfortable but tolerable
  3. severe, can only barely tolerate The higher the score, the more severe the anxiety symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, 3 months after surgery
  The PSQI contains 19 self-rated entries and 5 other rated entries, but only 19 self-rated entries participate in the score. The entries are divided into seven components, each scored on a 0-3 scale, with an overall score ranging from 0-21.
Blood immune inflammation indicators | Baseline
  such as interleukin-1β (IL-1β), IL-2, IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), interferon-γ (IFN-γ), C-reactive protein (CRP), calcitonin gene-related peptide (CGRP), neurofilament light chain (sNfL), glial fibrillary acidic protein (sGFAP).
PBC asscoated adverse reactions | 24 hours after surgery, 3 months after surgery
  such as hypoesthesia (numbness of the face and tongue), decreased corneal reflexes, dry eye, double vision, masseter weakness, oral herpes simplex